CLINICAL TRIAL: NCT06040684
Title: Development of Antibodies Against Transplant Kidney After Infection
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: INT-01-HLATX-Kidney; 15/RVO-FNOs/2018 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2018-05-23; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Acute Infection; Kidney Failure
Keywords: kidney transplant; HLA antibodies; acute infection
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Antibodies in blood samples (excessive material remaining after performing all necessary standard diagnostic tests) will be analyzed upon admission and then in 5 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Level of antibodies in kidney transplant recipients: Patients with kidney transplant with a severe acute infection will be enrolled in the study. Levels of antibodies in these patients will be analyzed.
  Interventions: Diagnostic Test: Level of antibodies

INTERVENTIONS:
Diagnostic Test: Level of antibodies — The level of antibodies against transplanted kidney in patients with a severe acute infection will be measured upon admission and then in 5 weeks.

SUMMARY:
Kidney transplantation is the best method of renal replacement in patients with irreversible renal failure. One of the biggest problems today is premature loss of function of the transplanted kidney. This occurs most often on the basis of chronic humoral rejection. This is the immune response to the kidney, in which the specific antibodies play a crucial role (both against the HLA and the non-HLA system).

The aim of this study is to analyze one of the situations where the production of antibodies can begin to occur. This is a serious acute infection (bacterial, viral, or fungal), where it is necessary to significantly reduce doses of immunosuppressives. At the time of reduced immunosuppression, the immune system can recognize the transplanted kidney as foreign to the human body and begin to fight against it.

In this study, the investigators will monitor antibodies against the transplanted kidney in patients with severe acute infection. A serious infection in this study is one that requires acute hospitalization and reduced doses of immunosuppressive drugs. The researchers will measure the antibodies in the blood upon admission and then in 5 weeks.

DETAILED DESCRIPTION:
Kidney transplantation significantly improves the prognosis and quality of life of patients with irreversible renal failure (end-stage kidney disease), requiring hemodialysis or peritoneal dialysis. The length of the function of the transplanted kidney depends on a number of factors. One of the most significant deterioration factors and subsequent graft function failure, in the long run, is the production of antibodies against HLA as well as transplant antigens that lead to acute or chronic humoral rejection. Chronic humoral rejection leading to transplant glomerulopathy is the most common cause of loss of function of the transplanted kidney. Treatment interventions in this area are still ineffective.

In spite of immunosuppressive therapy, some patients develop anti-transplant antibodies (both against HLA and non-HLA antibody molecules) even with stable graft function. However, these patients have an increased risk of losing their function due to chronic humoral rejection. The HLA-DR and HLA-DQ molecules have the greatest immunogenicity.

Patients after kidney transplantation may have many complications. Both surgical (vascular anastomoses stenoses, wound healing problems, graft vascular thromboses, lymphocele, urinary leakage) and non-surgical, some of which are immune-compromised (rejection) and others, result from the mechanism of action of immunosuppressive preparations (infections, cardiovascular effects). Amongst potentially life-threatening conditions include acute infections. Immunosuppressed infections have their own specifics. In addition to the increased risk of infections; also a different spectrum of possible originators is known. It is also possible to encounter opportunistic infections - pneumocystis, cytomegalovirus, polyomavirus infections. Another specific feature is often a different course of infection - patients may not have significantly expressed clinical or laboratory findings and may progress rapidly. For these reasons, physicians are often forced to significantly reduce immunosuppression rates in patients with acute infection, despite the increased risk of developing rejection. This situation increases the risk of initiation by both cell-mediated rejection and antibody-mediated rejection. Signs of rejection are very nonspecific and the only diagnostic method is graft biopsy. Previous studies have shown that the production of antibodies to the transplanted kidney is preceded by clinical signs of deterioration in graft function over weeks to months. Patients included in the study according to the criteria will be examined for the presence of HLA antibodies and non-HLA on admission (within 48 hours of admission) and 5 weeks after the first sample method LUMINEX xMAP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over.
* A kidney transplant patient - from a living donor or from a cadaveric donor (donor after circulatory or brain death). The patient will be included after 1st transplant and possible retransplantation.
* The patient is hospitalized or newly admitted to the FN Ostrava internal clinic for acute infection + requires the reduction of immunosuppressive therapy (dose reduction or discontinuation of any of the maintenance immunosuppressive preparations - tacrolimus, cyclosporin A, sirolimus, everolimus, azathioprine, mycophenolate).
* Acute infection (to be admitted to an internal clinic - determine the time of admission or the time of the first symptom of infection in the already hospitalized) occurred at least more than 48 hours after transplantation (from reperfusion time) and a maximum of 10 years after transplantation.
* The patient did not receive intravenous immunoglobulins within the last 24 hours prior to first sampling.
* This is not a pregnant woman.

Exclusion Criteria:

* Patient's death before the 2nd blood sampling.
* The patient condition was conclusively determined as something other than acute infection (acute rejection episode, acute pancreatitis, malignant tumor, ...). Unfamiliarity with localization of the infection or its origin, assuming an infectious etiology, is NOT an exclusion criterion.
* The patient was graftectomized - removal of the transplanted kidney, between the 1st and 2nd antibody determination.
* Detection of pregnancy when the term of conception is calculated before the 2nd antibody count.
* One or more transfusions of the erythrocytes or plasma between the 1st and 2nd measurements were administered to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients with acute infection (viral, bacterial or fungal) requiring acute inpatient care
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Production of HLA and nonHLA antibodies - Luminex | 42 months
  Screening for HLA and nonHLA antibodies by Luminex. The test result will be positive (MFI - mean fluorescence intensity above 300) or negative.

SECONDARY OUTCOMES:
Analysis of antibody formation according to age | 42 months
  The formation of antibodies will be analysed according to the age of the patients in years.
Analysis of antibody formation according to time from transplantation | 42 months
  The formation of antibodies will be analysed according to the time from transplantation in months.
Creatinine value | 42 months
  The baseline kidney function will be assessed (according to the KDIGO organization) The kidney will be classified as a normal function, 1st, 2nd, 3rd according to the creatinine value).
Input Inflammatory Parameters - CRP (C-reactive protein) | 42 months
  The input inflammatory parameters will be assessed (CRP (mg/l).
Input Inflammatory Parameters - IL-6 (Interleukin-6) | 42 months
  The input inflammatory parameters will be assessed (IL-6 (ng/l).
Number of HLA mismatches during transplant (0-6) | 42 months
  The number of HLA mismatches during transplant (0-6) will be recorded.
Length of immunosuppression reduction | 42 months
  The length of immunosuppression reduction will be analysed in 3 categories - up to 5 days, 5-10 days and over 10 days.
Delayed graft function after transplantation | 42 months
  The delayed graft function after transplantation will be assessed in 2 categories - YES / NO -as a need for haemodialysis in the first week after transplantation.
Long-term graft function | 42 months
  The long-term graft function will be assessed by the last early graft function (eGF) in ml / sec- 3 categories - normal function, G1-2 and G3-5 by KDIGO.
Type of infection | 42 months
  The type of infection observed in the patients will be assessed and recorded - urinary, respiratory, other - determined by the doctor when the patient is discharged.
Presence of antibodies | 42 months
  The presence of antibodies (YES/NO) will be determined in patients using the LUMINEX method - antibody value using MFI - mean fluorescence intensity.
EGF value | 42 months
  The function of the transplanted kidney will be assessed at 6 months (+ -14 days) from the first measurement assessing the EGF value (ml/sec)
Proteinuria | 42 months
  The function of the transplanted kidney will be assessed at 6 months (+ -14 days) from the first measurement assessing the proteinuria (g/l)

CONTACTS AND LOCATIONS:
Overall Officials: Zdeněk Lys, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make individual participant data available to other researchers.